CLINICAL TRIAL: NCT05196828
Title: Open-label Extension Study to Evaluate Longer-Duration Response to the NTX100 Neuromodulation System for Patients With Medication-Refractory Primary Restless Legs Syndrome (RLS)
Brief Title: Extension Study Evaluating NTX100 Neuromodulation System for Medication-Refractory Primary RLS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Noctrix Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT-05
Record Dates: First submitted 2021-12-31; First posted 2022-01-19 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Restless Legs Syndrome
MeSH Terms: conditions — Restless Legs Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Arm 1 - Direct Roll-Over Extension (Active Comparator): 24-wks of Active neurostimulation - Noninvasive peripheral nerve stimulation device programmed to deliver active stimulation; followed by 8-wks of No Intervention
  Interventions: Device: NTX100 Neuromodulation System
- Arm 2 - Control Group (No Intervention): 24-wks of No Intervention

INTERVENTIONS:
Device: NTX100 Neuromodulation System — Active Noninvasive peripheral nerve stimulation device programmed to active mode
  Arms: Arm 1 - Direct Roll-Over Extension

SUMMARY:
Multi-center, prospective open-label extension study of noninvasive peripheral nerve stimulation (NPNS) with the NTX100 Neuromodulation System for patients with medication-refractory moderate- severe primary RLS

DETAILED DESCRIPTION:
This is an extension study only inviting subjects who have previously completed the RESTFUL Study (NCT04874155).

Each study subject is enrolled into one of the following Arms:

Arm 1 (Direct Roll-Over Extension): 24-week open-label NPNS followed by 8-weeks of no treatment, no delay after completion of the RESTFUL Study

Arm 2 (Control Group): 24-weeks of no treatment

ELIGIBILITY:
Inclusion Criteria:

1. Subject previously completed the RESTFUL Study (NCT04874155).
2. Subject has signed a valid, Institutional Review Board-approved informed consent form, can understand the requirements of the study and instructions for device usage, and can converse in English.
3. [applicable to Arm 1 only] Subject agrees to not change dosage or schedule of any medications that are known to impact RLS symptoms during the study, including RLS medications, antidepressants, sleep medications, or sedative antihistamines.

Exclusion Criteria:

1. [applicable to Arm 1 only] Subject has active medical device implant anywhere in the body (including but not limited to pacemakers, spinal cord stimulators, deep brain stimulators) or metal implant at the site of study device electrode application.
2. [applicable to Arm 1 only] Subject has been diagnosed with one of the following conditions:

   * Epilepsy or other seizure disorder Current, active or acute or chronic infection other than common cold [and except for acute infections with mild symptoms]
   * A malignancy within the past 5 years (not including basal or squamous cell skin cancer)
   * Stage 4-5 chronic kidney disease or renal failure
   * Severe movement disorder symptoms (Parkinson's disease, Huntington's disease, dyskinesia, dystonia)
   * Deep vein thrombosis
   * Multiple sclerosis
3. Subject has moderate or severe cognitive disorder or mental illness.
4. [applicable to Arm 1 only] Subject has known allergy to device materials, electrode gel, polyurethane foam, or lycra (or severe previous reaction to medical adhesives or bandages).
5. [applicable to Arm 1 only] Subject has severe edema affecting lower legs.
6. [applicable to Arm 1 only] Subject has any of the following at or near the location of device application.

   * Acute injury
   * Cellulitis
   * Open sores
   * Other skin condition
7. [applicable to Arm 1 only] Subject is on dialysis or anticipated to start dialysis while participating in the study.
8. [applicable to Arm 1 only] Subject has received another investigational device or drug within 30 days before study entry, is planning to receive another investigational device or drug during the study, or is planning to change RLS medications during the study.
9. Subject is unable or unwilling to comply with study requirements.
10. [applicable to Arm 1 only] Subject is pregnant or trying to become pregnant.
11. Subject has a medical condition not listed above that may affect validity of the study as determined by the investigator.
12. [applicable to Arm 1 only] Subject has a medical condition not listed above that may put the subject at risk as determined by the investigator.
13. Subject was unwilling or unable to follow instructions in the RESTFUL Study, including missing 2 or more follow-up evaluations.
14. [applicable to Arm 1 only] Subject failed to properly operate the investigational devices during Weeks 5-8 of the RESTFUL Study.
15. [applicable to Arm 1 only] Subject experienced a significantly higher than expected rate of device malfunctions in the RESTFUL Study, such that the malfunctions appeared to be directly related to the subject's pattern of use.

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2022-09-27 (Actual); Study Completion 2022-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan D Charlesworth, PhD, Study Director — Noctrix Health, Inc.
Locations (7):
- United States (7):
  - California Center for Sleep Disorders, San Leandro, California
  - Delta Waves, Inc., Colorado Springs, Colorado
  - Neurotrials Research, Atlanta, Georgia
  - Clayton Sleep Institute, St Louis, Missouri
  - Ohio Sleep Medicine Institute, Dublin, Ohio
  - Bogan Sleep Consultants, LLC, Columbia, South Carolina
  - FutureSearch Trials of Neurology, Austin, Texas

REFERENCES:
- [Derived] Roy A, Ojile J, Kram J, Olin J, Rosenberg R, Hudson JD, Bogan RK, Charlesworth JD. Long-term efficacy and safety of tonic motor activation for treatment of medication-refractory restless legs syndrome: A 24-Week Open-Label Extension Study. Sleep. 2023 Oct 11;46(10):zsad188. doi: 10.1093/sleep/zsad188. PMID 37439365

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the parent study (CT-04, RESTFUL Study). The CT-04 study enrolled 133 subjects, 126 of which completed the study. These 126 subjects were invited to participate in the CT-05 Extension study but 23 were not enrolled (7 not reachable, 12 did not consent, 1 was ineligible and 3 were unable to enroll due to a site not yet active.). This left 103 subjects that were consented and enrolled in CT-05, the Extension study.
Period: Overall Study
Arm/Group | Arm 1 - Direct Roll-Over Extension | Arm 2 - Control Group
Started | 44 | 59
Completed | 41 | 55
Not Completed | 3 | 4
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lost to Follow-up | 0 | 4
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 - Direct Roll-Over Extension | Arm 2 - Control Group | Total
Number analyzed (Participants) | 44 | 59 | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.7 (11.65) | 57.5 (11.85) | 57.6 (11.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 32 | 58
  Male | 18 | 27 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 7
  Not Hispanic or Latino | 40 | 52 | 92
  Unknown or Not Reported | 0 | 4 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 40 | 52 | 92
  More than one race | 4 | 3 | 7
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects for Which the Clinician Reported "Much Improved" or "Very Much Improved" on the Clinical Global Impressions-Improvement (CGI-I) Scale in Treatment Group (Arm 1) Relative to Baseline.
Description: Responder rate is defined as the proportion of responses of "Much Improved" or "Very Much Improved" relative to baseline on the investigator-rated 7-point CGI-I scale. The outcomes were also evaluated as Treatment Group (Arm 1) at 24 weeks related to Control Group (Arm 2) at 24 weeks. The primary outcome, however, is the measure relative to baseline.
Time Frame: Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 - Direct Roll-Over Extension | Arm 2 - Control Group
Number analyzed (Participants) | 44 | 59
Participants | 32 | 8

2. Secondary Outcome: Number of Subjects That Report "Much Improved" or "Very Much Improved" on the Patient Global Impressions-Improvement (PGI-I) Scale in the Treatment Group (Arm 1) Relative to Baseline.
Description: Responder rate is defined as the proportion of responses "Much Improved" or "Very Much Improved" on the Patient Global Impressions-Improvement (PGI-I) Scale in the Treatment Group (Arm 1) Relative to Baseline. Note that the Responder Rate was be calculated relative to baseline for the endpoint but was also be calculated relative to the value for the control group at Week 24.
Time Frame: Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 - Direct Roll-Over Extension | Arm 2 - Control Group
Number analyzed (Participants) | 44 | 59
Participants | 33 | 12

3. Secondary Outcome: Mean Change From Baseline in International Restless Legs Syndrome Study Group Rating Scale (IRLS) Score in Arm 1
Description: IRLS is a participant-rated questionnaire that rates RLS severity from 0-40, where 40 is the most severe. Note that the IRLS score was calculated relative to baseline for the endpoint but was also be calculated relative to the value for the control group at Week 24.
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1 - Direct Roll-Over Extension | Arm 2 - Control Group
Number analyzed (Participants) | 44 | 59
score on a scale | -11.3 (8.43) | -5.4 (6.70)

4. Secondary Outcome: Mean Change From Baseline in Medical Outcomes Study Sleep Problems Index II (MOS-II) Score in Arm 1
Description: MOS-II is a subscale of the participant-rated MOS questionnaire that measures subjective sleep quality. The MOS-I (6-items) and MOS-II (9-items) are the two validated subscales of the 12-item MOS Sleep Scale. Both are scored from 0 to 100, where 100 corresponds to the worst possible sleep problems and 0 corresponds to no sleep problems. See https://labs.dgsom.ucla.edu/hays/files/view/docs/surveys/sleep/sleepman-112603.pdf for more information.
  Note that the mean MOS-II score was calculated relative to baseline for the endpoint but was also be calculated relative to the value for the control group at Week 24.
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1 - Direct Roll-Over Extension | Arm 2 - Control Group
Number analyzed (Participants) | 44 | 59
score on a scale | -17.2 (18.81) | -6.4 (15.18)

5. Secondary Outcome: Mean Change From Baseline in Medical Outcomes Study Sleep Problems Index I (MOS-I) Score in Arm 1
Description: MOS-I is a subscale of the participant-rated MOS questionnaire that measures subjective sleep quality. The MOS-I (6-items) and MOS-II (9-items) are the two validated subscales of the 12-item MOS Sleep Scale. Both are scored from 0 to 100, where 100 corresponds to the worst possible sleep problems and 0 corresponds to no sleep problems. See https://labs.dgsom.ucla.edu/hays/files/view/docs/surveys/sleep/sleepman-112603.pdf for more information. Note that the outcome is measured relative to baseline but also relative to the Arm 2 (control group) at 24 weeks.
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1 - Direct Roll-Over Extension | Arm 2 - Control Group
Number analyzed (Participants) | 44 | 59
score on a scale | -15.8 (19.21) | -5.7 (15.48)

6. Secondary Outcome: Days Per Week of RLS Symptoms Based on Question #7 in the International Restless Legs Syndrome Study Group Rating Scale (IRLS) Score in Arm 1
Description: The International Restless Legs Syndrome (IRLS) Question #7 is a participant-rated question that measures the frequency of RLS symptoms in terms of days per week.
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: Days/Week
Arm/Group | Arm 1 - Direct Roll-Over Extension | Arm 2 - Control Group
Number analyzed (Participants) | 44 | 59
Days/Week | -1.50 (1.34) | -0.41 (0.91)

ADVERSE EVENTS:
Time Frame: Up to 32 weeks.
Description: Descriptive analyses of adverse events for both study arms, classified and tabulated by seriousness, relationship to the device, and severity.
Groups:
- Arm 1: Treatment Group
- Arm 2: Control Group
Arm/Group | Arm 1 | Arm 2
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/44
Other Adverse Events (participants affected / at risk) | 10/44 | 3/44
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=44) | Arm 2 (N=44)
Discomfort (Skin and subcutaneous tissue disorders) | 10 (10) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-11-24): https://cdn.clinicaltrials.gov/large-docs/28/NCT05196828/Prot_003.pdf
  • Statistical Analysis Plan (2023-03-10): https://cdn.clinicaltrials.gov/large-docs/28/NCT05196828/SAP_004.pdf